CLINICAL TRIAL: NCT03341780
Title: Standard Amblyopia Therapy in Adult Amblyopes
Status: Completed | Type: Observational
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: SoutherCCO
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: amblyopia therapy — Any of the following amblyopia training activities may be employed during patching: board games, card games, coloring in O's, comic books, craft projects, crossword puzzles, dot-to-dot patterns, drawing, hammering nails, jacks, jigsaw puzzles, lego and other blocks, marbles, mazes, peg-board activities, perceptual materials, pickup sticks, reading, sewing, shooting games, stringing beads, throwing or hitting games, tracing, and video or computer games.

SUMMARY:
Amblyopia is characterized by a reduction in visual acuity, contrast sensitivity, and binocular visual functions. The two main causes of amblyopia are anisometropia and strabismus which alter the synaptic connections between neurons along the visual pathway. Current treatment for amblyopia has indicated that the younger the amblyope, the greater the effect of treatment. The purpose of this study is to determine if standard amblyopia treatment improved visual acuity in adult amblyopes.

DETAILED DESCRIPTION:
Functional amblyopia is an optically uncorrectable decrease in visual acuity, i.e., spatial resolution, with no apparent pathological or morphological cause. There are several etiological origins for amblyopia in the human population; anisometropia and strabismus are the two most prevalent etiological factors. Anisometropic amblyopia is a decrease in visual acuity (spatial resolution) that is the result of a large difference in refractive error between the two eyes. Strabismic amblyopia is characterized by an eye misalignment early in life which is associated with a decrease in visual acuity.

The initial site of the defect in amblyopia is the primary visual cortex. The amblyopic eye is placed at a competitive disadvantage to the nonamblyopic eye which results in a reduction in the synapses or cells responding to the amblyopic eye. The conditions associated with amblyopia must be present prior to the end of the critical period of neural development for amblyopia to develop. The neurophysiological systems of anisometropic and strabismic monkeys have differences in the distributions of binocular cortical cells. Anisometropic amblyopic monkeys only exhibit binocular cells that are tuned to low spatial frequencies. If a neuron has a high spatial resolution, it is unlikely that the neuron will be binocular. However, strabismic amblyopic monkeys exhibit few binocular cells and, moreover, there does not appear to be a spatial frequency dependent distribution of these binocular cells. The strabismic subjects typically displayed few binocular cells, regardless of the spatial frequency tuning of the cell.

If the amblyopic eye is compared to the nonamblyopic eye, two important differences are noted. First, the amblyopic eye has a lower contrast sensitivity at high spatial frequencies (and sometimes at all spatial frequencies) than the nonamblyopic eye. This also results in a decrease in visual acuity for the amblyopic eye. Second, the amblyopic eye demonstrates a longer latency for neural transmission than the nonamblyopic eye.

There is very little published on adult amblyopia therapy. This is because clinicians initially believed that amblyopia could not be treated after the end of the critical period. The prevailing theory was that the synaptic contacts between cells could only be modified during the critical period. In children, the majority of the improvement in acuity (80%) takes place in the first 6 weeks of therapy. There is a direct relationship between the hours of patching and the improvement in acuity. Most of the improvement in acuity occurs after the first 100 hours of patching.

There is a linear dose-response function for amblyopia treatment. The logMAR acuity increases 0.1 log unit or 1 chart line per 120 hours of patching. The response does not differ between the types of amblyopia. It has also been demonstrated that there is only a minimal benefit to patching more than 2 hours/day.

In a Pediatric Eye Disease Investigator Group (PEDIG) study, 189 amblyopic children were treated with 2 hours of patching per day. The amblyopic eye acuities ranged from 20/40 - 20/80 before treatment. The average improvement in acuity after 4 months of treatment was 0.24 logMAR (2.4 lines improvement on a logMAR chart). Another study used amblyopes with poorer acuity (20/100 - 20/400 before therapy). After 4 months of patching, the average increase in acuity was 0.48 logMAR (or an increase of 4.8 lines on a logMAR chart). The average acuity went from 20/250 (i.e., 1.10 logMAR) before treatment to 20/63 (i.e., 0.50 logMAR) after treatment. The results were the same for anisometropic amblyopes and strabismic amblyopes. In another study with amblyopes with starting acuity worse than 20/100, the improvement was 3.7 ± 2.5 logMAR chart lines of acuity.

Recent studies have suggested that adult amblyopia can be treated with non-standard therapy. Patching combined with active, near, threshold-training tasks and continuous feedback is employed in these studies. These studies indicate that amblyopia can be treated after the critical period ends. It is suggested that these perceptual learning tasks improve performance in the amblyopic eye by decreasing neural noise. Standard amblyopia therapy typically employed in children has not been investigated in adult amblyopes. The purpose of this study is to use standard amblyopic therapy to determine if there is an enhancement in visual performance in the amblyopic eye of adults.

ELIGIBILITY:
Inclusion Criteria:

* Amblyopic patients with acuities between 20/40 (0.30 logMAR) and 20/400 (1.30 logMAR).
* All subjects will be over the age of 18.
* Prior amblyopia therapy is not an exclusion criteria.
* Subjects will be recruited from the College community and University Eye Clinic.

Exclusion Criteria:

* A significant cataract that affects vision.
* Glaucoma, diabetes, uncontrolled high blood pressure.
* Other ocular or systemic diseases that will affect visual acuity.
* The inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the College community and University Eye Clinic. An announcement will be made to the College community and volunteers accepted.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

PRIMARY OUTCOMES:
visual acuity | 24 weeks
  LogMAR acuity will be measured with the eETDRS chart

CONTACTS AND LOCATIONS:
Overall Officials: William Ridder, OD, PhD, Principal Investigator — Southern California College of Optometry at Marshall B. Ketchum University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] von Noorden GK. Amblyopia: a multidisciplinary approach. Proctor lecture. Invest Ophthalmol Vis Sci. 1985 Dec;26(12):1704-16. PMID 3934105
- [Background] Michaels DD. Visual optics and refraction: a clinical approach. St Louis, MO: C.V. Mosby Co.; 1980.
- [Background] Crawford ML, Blake R, Cool SJ, von Noorden GK. Physiological consequences of unilateral and bilateral eye closure in macaque monkeys: some further observations. Brain Res. 1975 Jan 24;84(1):150-4. doi: 10.1016/0006-8993(75)90809-4. No abstract available. PMID 1111823
- [Background] Hubel DH, Wiesel TN, LeVay S. Plasticity of ocular dominance columns in monkey striate cortex. Philos Trans R Soc Lond B Biol Sci. 1977 Apr 26;278(961):377-409. doi: 10.1098/rstb.1977.0050. No abstract available. PMID 19791
- [Background] Stewart CE, Moseley MJ, Stephens DA, Fielder AR. Treatment dose-response in amblyopia therapy: the Monitored Occlusion Treatment of Amblyopia Study (MOTAS). Invest Ophthalmol Vis Sci. 2004 Sep;45(9):3048-54. doi: 10.1167/iovs.04-0250. PMID 15326120
- [Background] Repka MX, Beck RW, Holmes JM, Birch EE, Chandler DL, Cotter SA, Hertle RW, Kraker RT, Moke PS, Quinn GE, Scheiman MM; Pediatric Eye Disease Investigator Group. A randomized trial of patching regimens for treatment of moderate amblyopia in children. Arch Ophthalmol. 2003 May;121(5):603-11. doi: 10.1001/archopht.121.5.603. PMID 12742836
- [Background] Holmes JM, Kraker RT, Beck RW, Birch EE, Cotter SA, Everett DF, Hertle RW, Quinn GE, Repka MX, Scheiman MM, Wallace DK; Pediatric Eye Disease Investigator Group. A randomized trial of prescribed patching regimens for treatment of severe amblyopia in children. Ophthalmology. 2003 Nov;110(11):2075-87. doi: 10.1016/j.ophtha.2003.08.001. PMID 14597512
- [Background] Holmes JM, Edwards AR, Beck RW, Arnold RW, Johnson DA, Klimek DL, Kraker RT, Lee KA, Lyon DW, Nosel ER, Repka MX, Sala NA, Silbert DI, Tamkins S; Pediatric Eye Disease Investigator Group. A randomized pilot study of near activities versus non-near activities during patching therapy for amblyopia. J AAPOS. 2005 Apr;9(2):129-36. doi: 10.1016/j.jaapos.2004.12.014. PMID 15838439
- [Background] Holmes JM, Lazar EL, Melia BM, Astle WF, Dagi LR, Donahue SP, Frazier MG, Hertle RW, Repka MX, Quinn GE, Weise KK; Pediatric Eye Disease Investigator Group. Effect of age on response to amblyopia treatment in children. Arch Ophthalmol. 2011 Nov;129(11):1451-7. doi: 10.1001/archophthalmol.2011.179. Epub 2011 Jul 11. PMID 21746970
- [Background] Levi DM, Li RW. Perceptual learning as a potential treatment for amblyopia: a mini-review. Vision Res. 2009 Oct;49(21):2535-49. doi: 10.1016/j.visres.2009.02.010. Epub 2009 Feb 27. PMID 19250947
- [Background] Levi DM, Li RW. Improving the performance of the amblyopic visual system. Philos Trans R Soc Lond B Biol Sci. 2009 Feb 12;364(1515):399-407. doi: 10.1098/rstb.2008.0203. PMID 19008199
- [Background] Ridder WH 3rd, Rouse MW. Predicting potential acuities in amblyopes: predicting post-therapy acuity in amblyopes. Doc Ophthalmol. 2007 May;114(3):135-45. doi: 10.1007/s10633-007-9048-y. Epub 2007 Feb 20. PMID 17310345